CLINICAL TRIAL: NCT03819504
Title: STereotactic Ablative Radiosurgery of Recurrent Ventricular Tachycardia in Structural Heart Disease
Brief Title: Stereotactic Non-invasive Ablation of Ventricular Tachycardia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in the design of the study
Sponsor: University Hospital Ostrava (Other)
Collaborators: Institute for Clinical and Experimental Medicine (Other Government); Hospital Podlesi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR-VT; NV19-02-00212 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Ventricular Tachycardia
Keywords: Structural Heart Disease; Ventricular Tachycardia; Substrate Ablation; Stereotactic Radiosurgery; Functional Radiosurgery; 4D navigation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-D navigated stereotactic radiosurgical ablation (Experimental): Patients with structural heart disease and sustained monomorphic ventricular tachycardia/tachycardias will undergo 4-D navigated stereotactic radiosurgical ablation
  Interventions: Procedure: 4-D navigated stereotactic radio surgical ablation

INTERVENTIONS:
Procedure: 4-D navigated stereotactic radio surgical ablation — 4-D navigated stereotactic radio surgical ablation will be performed in patients with structural heart disease and sustained monomorphic ventricular tachycardia/tachycardias

SUMMARY:
STereotactic Ablative Radiosurgery of recurrent Ventricular Tachycardia in structural heart disease (STAR-VT).

DETAILED DESCRIPTION:
The goal of this project is to evaluate feasibility and safety/toxicity of elimination of ventricular tachycardia (VT) associated with structural heart disease by noninvasive strategy, stereotactic radiosurgical ablation in an indication of bail-out procedure after failed catheter ablation. The arrhythmogenic substrate will be identified by imaging techniques and functionally by electroanatomic mapping and pacing. The recipients of stereotactic surgery will be patients after 2 unsuccessful catheter ablations for monomorphic VTs (one of the procedures will be performed in an expert center). The target volume for stereotactic radiosurgical ablation (single dose of 25 Gy) will be a critical region of the substrate defined by a combination of imaging and functional methods with an export of the merged image-electroanatomical map into the radiosurgery planning console. Primary endpoints will be a reduction of the burden of sustained VT, time to death or arrhythmic storm or appropriate therapy with implantable cardioverter-defibrillator (ICD) for isolated VT and/or time do development of radiation toxicity (both acute and late).

ELIGIBILITY:
Inclusion Criteria:

* Patients with structural heart disease (ischemic and non-ischemic cardiomyopathy, previous surgery for congenital heart disease)
* Implanted ICD or CRT-D (cardiac resynchronization therapy defibrillator)
* Prior ≥1 catheter ablation procedure for monomorphic VT
* VT recurrence early (<12 months) after the last ablation with at least 2 episodes of recurrent VT, including 1 episode while on amiodarone (if not contraindicated)
* Age ≥30 years
* Signed an IRB-approved (Institutional Review Board) written informed consent

Exclusion Criteria:

* Acute myocardial infarction or recent percutaneous coronary intervention (PCI) or cardiac surgery (<3 months)
* Primary electrical disease (channelopathy)
* Reversible cause of VT (e.g. drug-induced, intoxications, etc)
* Pregnancy or breastfeeding
* Chronic heart failure New York Heart Association (NYHA) Class IV
* Serious comorbidities with presumed life expectancy less than one year
* Significant peripheral artery disease precluding retrograde aortic mapping
* History of chest radiotherapy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change of sustained VT burden in three 3-month intervals | 50 months
  Change of sustained VT burden in three 3-month intervals will be assessed. For all arrhythmic events, a 90-day post-radiosurgery blanking period will be applicable.
Composite endpoint of (i) all-cause death, (ii) appropriate ICD therapy (both shock and antitachycardia pacing) for VT/VF (ventricular fibrillation) or (iii) sustained VT below the detection threshold | 50 months
  All-cause death, appropriate ICD therapy (both shock and antitachycardia pacing) for VT/VF (ventricular fibrillation) or sustained VT below the detection threshold will be observed for up to 50 months. For all arrhythmic events, a 90-day post-radiosurgery blanking period will be applicable.
3. Rate of acute (<3 months) and late radiation-induced events according to CTCAE 4.0. | 53 months
  The rate of acute (<3 months) and late radiation-induced events according to CTCAE 4.0 will be observed.

SECONDARY OUTCOMES:
Composite endpoint of all-cause death and appropriate ICD shock | 50 months
  The composite endpoint of all-cause death and appropriate ICD shock will be observed for the period of up to 50 months. For all arrhythmic events, a 90-day post-radiosurgery blanking period will be applicable.
Electric storm recurrence | 53 months
  The recurrence of electric storm will be observed. For all arrhythmic events, a 90-day post-radiosurgery blanking period will be applicable.
Cardiovascular hospitalisations | 53 months
  The hospitalisations due to cardiovascular indications will be observed.
Change in quality of life | 53 months
  Change in quality of life will be observed using the standardised EQ-5D (5-dimension) questionnaire. EQ-5D is a standardised instrument in the form of a questionnaire developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The quality of life is assessed in five dimensions, with three levels in each dimension. The higher score the patient achieves, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Cvek, Ass.Prof.,MD,Ing.,PhD, Study Chair — University Hospital Ostrava
Locations (3):
- Czechia (3):
  - Institute for Clinical and Experimental Medicine Prague, Prague, Central Bohemia
  - University Hospital Ostrava, Ostrava-Poruba, Czech Republic
  - Hospital Podlesí, Třinec, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not decided to share the individual participant data with other researchers.

REFERENCES:
- [Background] Connolly SJ, Hallstrom AP, Cappato R, Schron EB, Kuck KH, Zipes DP, Greene HL, Boczor S, Domanski M, Follmann D, Gent M, Roberts RS. Meta-analysis of the implantable cardioverter defibrillator secondary prevention trials. AVID, CASH and CIDS studies. Antiarrhythmics vs Implantable Defibrillator study. Cardiac Arrest Study Hamburg . Canadian Implantable Defibrillator Study. Eur Heart J. 2000 Dec;21(24):2071-8. doi: 10.1053/euhj.2000.2476. PMID 11102258
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Connolly SJ, Dorian P, Roberts RS, Gent M, Bailin S, Fain ES, Thorpe K, Champagne J, Talajic M, Coutu B, Gronefeld GC, Hohnloser SH; Optimal Pharmacological Therapy in Cardioverter Defibrillator Patients (OPTIC) Investigators. Comparison of beta-blockers, amiodarone plus beta-blockers, or sotalol for prevention of shocks from implantable cardioverter defibrillators: the OPTIC Study: a randomized trial. JAMA. 2006 Jan 11;295(2):165-71. doi: 10.1001/jama.295.2.165. PMID 16403928
- [Background] Moss AJ, Schuger C, Beck CA, Brown MW, Cannom DS, Daubert JP, Estes NA 3rd, Greenberg H, Hall WJ, Huang DT, Kautzner J, Klein H, McNitt S, Olshansky B, Shoda M, Wilber D, Zareba W; MADIT-RIT Trial Investigators. Reduction in inappropriate therapy and mortality through ICD programming. N Engl J Med. 2012 Dec 13;367(24):2275-83. doi: 10.1056/NEJMoa1211107. Epub 2012 Nov 6. PMID 23131066
- [Background] Mallidi J, Nadkarni GN, Berger RD, Calkins H, Nazarian S. Meta-analysis of catheter ablation as an adjunct to medical therapy for treatment of ventricular tachycardia in patients with structural heart disease. Heart Rhythm. 2011 Apr;8(4):503-10. doi: 10.1016/j.hrthm.2010.12.015. Epub 2010 Dec 13. PMID 21147263
- [Background] Sapp JL, Wells GA, Parkash R, Stevenson WG, Blier L, Sarrazin JF, Thibault B, Rivard L, Gula L, Leong-Sit P, Essebag V, Nery PB, Tung SK, Raymond JM, Sterns LD, Veenhuyzen GD, Healey JS, Redfearn D, Roux JF, Tang AS. Ventricular Tachycardia Ablation versus Escalation of Antiarrhythmic Drugs. N Engl J Med. 2016 Jul 14;375(2):111-21. doi: 10.1056/NEJMoa1513614. Epub 2016 May 5. PMID 27149033
- [Background] Aldhoon B, Wichterle D, Peichl P, Cihak R, Kautzner J. Outcomes of ventricular tachycardia ablation in patients with structural heart disease: The impact of electrical storm. PLoS One. 2017 Feb 10;12(2):e0171830. doi: 10.1371/journal.pone.0171830. eCollection 2017. PMID 28187168
- [Background] Raymond JM, Sacher F, Winslow R, Tedrow U, Stevenson WG. Catheter ablation for scar-related ventricular tachycardias. Curr Probl Cardiol. 2009 May;34(5):225-70. doi: 10.1016/j.cpcardiol.2009.01.002. PMID 19348944
- [Background] Kumar S, Baldinger SH, Romero J, Fujii A, Mahida SN, Tedrow UB, Stevenson WG. Substrate-Based Ablation Versus Ablation Guided by Activation and Entrainment Mapping for Ventricular Tachycardia: A Systematic Review and Meta-Analysis. J Cardiovasc Electrophysiol. 2016 Dec;27(12):1437-1447. doi: 10.1111/jce.13088. Epub 2016 Oct 6. PMID 27574120
- [Background] Jais P, Maury P, Khairy P, Sacher F, Nault I, Komatsu Y, Hocini M, Forclaz A, Jadidi AS, Weerasooryia R, Shah A, Derval N, Cochet H, Knecht S, Miyazaki S, Linton N, Rivard L, Wright M, Wilton SB, Scherr D, Pascale P, Roten L, Pederson M, Bordachar P, Laurent F, Kim SJ, Ritter P, Clementy J, Haissaguerre M. Elimination of local abnormal ventricular activities: a new end point for substrate modification in patients with scar-related ventricular tachycardia. Circulation. 2012 May 8;125(18):2184-96. doi: 10.1161/CIRCULATIONAHA.111.043216. Epub 2012 Apr 4. PMID 22492578
- [Background] Di Biase L, Santangeli P, Burkhardt DJ, Bai R, Mohanty P, Carbucicchio C, Dello Russo A, Casella M, Mohanty S, Pump A, Hongo R, Beheiry S, Pelargonio G, Santarelli P, Zucchetti M, Horton R, Sanchez JE, Elayi CS, Lakkireddy D, Tondo C, Natale A. Endo-epicardial homogenization of the scar versus limited substrate ablation for the treatment of electrical storms in patients with ischemic cardiomyopathy. J Am Coll Cardiol. 2012 Jul 10;60(2):132-41. doi: 10.1016/j.jacc.2012.03.044. PMID 22766340
- [Background] Tzou WS, Frankel DS, Hegeman T, Supple GE, Garcia FC, Santangeli P, Katz DF, Sauer WH, Marchlinski FE. Core isolation of critical arrhythmia elements for treatment of multiple scar-based ventricular tachycardias. Circ Arrhythm Electrophysiol. 2015 Apr;8(2):353-61. doi: 10.1161/CIRCEP.114.002310. Epub 2015 Feb 13. PMID 25681389
- [Background] Tung R, Michowitz Y, Yu R, Mathuria N, Vaseghi M, Buch E, Bradfield J, Fujimura O, Gima J, Discepolo W, Mandapati R, Shivkumar K. Epicardial ablation of ventricular tachycardia: an institutional experience of safety and efficacy. Heart Rhythm. 2013 Apr;10(4):490-8. doi: 10.1016/j.hrthm.2012.12.013. Epub 2012 Dec 11. PMID 23246598
- [Background] Tokuda M, Kojodjojo P, Tung S, Tedrow UB, Nof E, Inada K, Koplan BA, Michaud GF, John RM, Epstein LM, Stevenson WG. Acute failure of catheter ablation for ventricular tachycardia due to structural heart disease: causes and significance. J Am Heart Assoc. 2013 May 31;2(3):e000072. doi: 10.1161/JAHA.113.000072. PMID 23727700
- [Background] Loo BW Jr, Soltys SG, Wang L, Lo A, Fahimian BP, Iagaru A, Norton L, Shan X, Gardner E, Fogarty T, Maguire P, Al-Ahmad A, Zei P. Stereotactic ablative radiotherapy for the treatment of refractory cardiac ventricular arrhythmia. Circ Arrhythm Electrophysiol. 2015 Jun;8(3):748-50. doi: 10.1161/CIRCEP.115.002765. No abstract available. PMID 26082532
- [Background] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642
- [Background] Chang SD, Main W, Martin DP, Gibbs IC, Heilbrun MP. An analysis of the accuracy of the CyberKnife: a robotic frameless stereotactic radiosurgical system. Neurosurgery. 2003 Jan;52(1):140-6; discussion 146-7. doi: 10.1097/00006123-200301000-00018. PMID 12493111
- [Background] Fariselli L, Marras C, De Santis M, Marchetti M, Milanesi I, Broggi G. CyberKnife radiosurgery as a first treatment for idiopathic trigeminal neuralgia. Neurosurgery. 2009 Feb;64(2 Suppl):A96-101. doi: 10.1227/01.NEU.0000341714.55023.8F. PMID 19165081
- [Background] Jumeau R, Ozsahin M, Schwitter J, Vallet V, Duclos F, Zeverino M, Moeckli R, Pruvot E, Bourhis J. Rescue procedure for an electrical storm using robotic non-invasive cardiac radio-ablation. Radiother Oncol. 2018 Aug;128(2):189-191. doi: 10.1016/j.radonc.2018.04.025. Epub 2018 May 9. PMID 29753550
- [Background] Regis J, Tuleasca C, Resseguier N, Carron R, Donnet A, Gaudart J, Levivier M. Long-term safety and efficacy of Gamma Knife surgery in classical trigeminal neuralgia: a 497-patient historical cohort study. J Neurosurg. 2016 Apr;124(4):1079-87. doi: 10.3171/2015.2.JNS142144. Epub 2015 Sep 4. PMID 26339857